CLINICAL TRIAL: NCT02883738
Title: Evaluation the Effect of Muscle Functional Electrical Stimulation in the Upper Limb Tremor Invalidating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 8188
Record Dates: First submitted 2016-08-09; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Upper Limb Tremor Invalidating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- upper limb tremor (Experimental)
  Interventions: Other: tremor

INTERVENTIONS:
Other: tremor — evaluation of the intensity of the tremor

SUMMARY:
The main objective of this study is to identify the superficial muscle groups involved in gene-related tremor and assess the reduction in the intensity of the tremor after transient electrical stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Subject with disabling tremor of upper limb
* Subject with essential tremor action and / or lesion

Exclusion Criteria:

* Subject with drug tremor
* Subject presenting an exaggerated physiological tremor
* Subject with isolated resting tremor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
evaluation of the intensity of tremor by measuring the hand moving speed (mm / s) | at day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Gui de Chauliac Hospital, Montpellier, France